CLINICAL TRIAL: NCT05069831
Title: JAK Inhibition in Food Allergy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Scott Sicherer, Professor, Pediatrics, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 21-0781
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Food Allergy
Keywords: Food Allergy; JAK; JAK Inhibitor; Abrocitinib; Immunoglobulin E
MeSH Terms: conditions — Food Hypersensitivity | interventions — abrocitinib

STUDY DESIGN:
Intervention Model Description: This is a single center, blinded, randomized pilot study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abrocitinib 100mg (Active Comparator): This arm will receive 100mg of the study drug
  Interventions: Drug: Abrocitinib
- Abrocitinib 200mg (Active Comparator): This arm will receive 200mg of the study drug
  Interventions: Drug: Abrocitinib

INTERVENTIONS:
Drug: Abrocitinib — Abrocitinib daily for 4 months

SUMMARY:
This study will assess the role for an oral targeted medication, abrocitinib, as a new treatment option for food allergy patients that would avoid injections. Abrocitinib, which has successfully completed phase three trials for atopic dermatitis, could serve as a single therapy for two conditions in many patients with multiple atopic conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 50 years old
* Participant must be able to understand and perform informed consent.
* IgE-mediated food allergy to at least one of the following foods as defined by (regarding at least one of the foods):

  ° Foods: peanut, cashew, walnut, hazelnut, sesame, cod, and/or shrimp, history of an acute allergic reaction (urticaria, angioedema, cough, wheeze, and/or repetitive vomiting within an hour of ingestion, and history of positive skin or serum IgE test, and current strict avoidance of the food, and current possession of physician-prescribed self-injectable epinephrine, and skin test wheal 5 mm or greater average diameter
* Current or past eczema.
* If female of childbearing potential, must have a negative pregnancy test (serum or urine) and agree to abstinence or acceptable contraception.
* Plan to remain in the Tri-State area during the trial for visits.
* Must agree to avoid prolonged exposure to the sun and not to use tanning booths, sunlamps, or other ultraviolet (UV) light sources during the study.
* If receiving concomitant medications for any reason other than AD, must be on a stable regimen, which is defined as not starting a new drug or changing dosage within 7 days or 5 half-lives (whichever is longer) prior to Day 1 and through the duration of the study.

Exclusion Criteria:

* Unwilling or unable to give written informed consent or comply with protocol.
* Unable to swallow pill.
* Use of dupilumab within 6 weeks of enrollment.
* Prior use or allergy to drugs related to abrocitinib (ruxolitinib, upadacitinib, etc).
* Use of any other biologic (monoclonal antibody) medication within 12 weeks or 5 half-lives of drug, if known.
* Allergy to any excipients within abrocitinib.
* Use of build-up environmental immunotherapy; any food oral immunotherapy;or systemic oral, IV or IM steroids including but not limited to- prednisone, methylprednisolone, prednisolone, solumedrol, solucortef, dexamethasone in the past 4 weeks or 5 half-lives of drug, if known.
* Use of CYP2C9 and CYP2C19 inducers (such as carbamazepine, norfluoxetine, etc.) within 5 half-lives of the inducer plus 14 days prior to the first dose of study intervention.
* Use of CYP2C9 and CYP2C19 inhibitors within 1 week of first dose of study intervention or within 5 half-lives (if known) of the inhibitor, whichever is longer.
* Unable to stop long-acting antihistamines within minimum wash out period required for SPTs at screening and site visits
* History of or significant risk factor(s) for cardiovascular disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
change in basophil activation | baseline and after 4 months of treatment
  change in basophil activation as measured by %CD63 AUC
change in skin prick test | baseline and after 4 months of treatment
  change in skin prick test size after four months of therapy.

SECONDARY OUTCOMES:
change in antigen-specific T-cell | baseline and after 4 months of treatment
  change in antigen-specific T-cell response
change in specific immunoglobulin E (sIgE) | baseline and after 4 months of treatment
  change in sIgE to allergic trigger food(s)
change in FENO | baseline and after 4 months of treatment
  Fractional Exhaled Nitric Oxide (FeNO) level

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sicherer, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Emma Guttman, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
data will be provided as a manuscript

REFERENCES:
- [Derived] Ghelli C, Costanzo G, Canonica GW, Heffler E, Paoletti G. New evidence in food allergies treatment. Curr Opin Allergy Clin Immunol. 2024 Aug 1;24(4):251-256. doi: 10.1097/ACI.0000000000000999. Epub 2024 May 30. PMID 38814736

DOCUMENTS (1):
  • Informed Consent Form (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT05069831/ICF_000.pdf